CLINICAL TRIAL: NCT03716531
Title: PACER (Pancreatic AdenoCarcinoma With Electron Intraoperative Radiation Therapy): A Phase II Study of Electron Beam Intraoperative Radiation Therapy Following Chemoradiation in Patients With Pancreatic Cancer With Vascular Involvement
Brief Title: Electron Beam Intraoperative Radiation Therapy Following Chemoradiation in Patients With Pancreatic Cancer With Vascular Involvement
Acronym: PACER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: IntraOp/Mobetron (Unknown)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-267
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- IORT (Experimental): * IORT will be administered as determined to be best practice by the treating radiation oncologist,
  * Electron beam intraoperative radiation therapy will occur in a hybrid operating room with a portable linear accelerator
  Interventions: Radiation: IORT

INTERVENTIONS:
Radiation: IORT — IORT works by delivering radiation therapy to the tumor while reducing the amount of healthy tissue exposed to the radiation therapy

SUMMARY:
This research study is studying an intervention as a possible treatment for pancreatic cancer.

DETAILED DESCRIPTION:
In this research study, the investigators are researching how well IORT during surgery works in treating pancreatic cancer after 3-6 months of chemotherapy and external radiation therapy. IORT works by delivering radiation therapy to the tumor while reducing the amount of healthy tissue exposed to the radiation therapy. The investigators believe that the administration of IORT after 3-6 months of chemotherapy will help to stop the cancer cells from growing.

The FDA (the U.S. Food and Drug Administration) has not approved IORT for this specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG Performance Status 0-1
* Previous completion of at least three (3) months of EITHER gemcitabine plus nab-paclitaxel OR FOLFIRINOX (5-fluorouracil, oxaliplatin, irinotecan and leucovorin)
* Previous completion of either stereotactic-body radiation therapy (SBRT) (minimum 24 Gy) or external beam irradiation (EBRT) (minimum 45 Gy)
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment is PERMITTED.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months after IORT.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after IORT. Women who are not of childbearing potential, i.e., who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of disease progression or distant metastases.
* Pregnant or lactating women
* Treatment for other invasive carcinomas within the last five years who are at greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* An active infection requiring systemic therapy
* Other serious medical conditions that the investigator feels might compromise study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
2 Year Overall Survival | 2 years
  Overall survival is defined as the time from IORT to death due to any cause, or is censored at the date of last follow-up, when applicable.

SECONDARY OUTCOMES:
Median Progression Free Survival | 2 years
  Progression-free survival is defined as the time from the date of IORT until the first evidence of local progression or distant metastasis (determined by imaging or biopsy) or death, and is censored at date of last follow-up when applicable.
Local Control | 2 years
  Local control is the absence of local failure, defined as evidence of growth or regrowth of the primary tumor and/or extension to regional lymph nodes that meets criteria for progressive disease beyond that present in pre-IORT imaging studies.
Adverse events associated with IORT | 2 years
  Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - University of California, Irvine, Irvine, California
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of North, Carolina Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No